CLINICAL TRIAL: NCT05450575
Title: A Prospective, Observational Study of Factors Affecting Blood Pressure and Blood Lipids After Treatment With Amosartan Q Tablet in Hypertension Patients With Dyslipidemia
Brief Title: An Observational Study to Evaluate Effectiveness and Safety of Amosartan Q Tablet
Status: Completed | Type: Observational
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: HM-AMOQ-OS-01
Record Dates: First submitted 2022-07-05; First posted 2022-07-08 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Hypertension; Dyslipidemia
Keywords: Amosartan; Hypertension; Dyslipidemia; Observational
MeSH Terms: conditions — Hypertension; Dyslipidemias

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- single arm, single group(No interventional): Observational
  Interventions: Drug: Amosartan Q tablet

INTERVENTIONS:
Drug: Amosartan Q tablet — Amlodipine, Losartan, Rosuvastatin
  Other Names: amosartan Q

SUMMARY:
This study was to evaluate the therapeutic effect and safety of amosartan Q tablet administration in adult patients with hypertension and dyslipidemia.

During the routine medical visit, Amosartan Q tablets were administered to patients in need of blood pressure/LDL-C control according to the investigator's judgment. In this study, effectiveness and safety information of treatment of Amosartan Q tablets was followed for 6 months (up to 12 months), and observation of the target patients was terminated after collecting relevant data.

As this study was a non-interventional observational study, all patients received prescriptions according to the routine treatment procedure, and there were no visits or procedures required according to the observational study protocol.

DETAILED DESCRIPTION:
This study was a multicenter, prospective, non-interventional, observational study of factors affecting blood pressure and blood lipids after treatment with Amosartan Q tablet in hypertension patients with dyslipidemia.

Data was collected from patients receiving routine treatment at hospitals in South Korea. Each patient visited the institution according to the protocol that designed the follow-up visits for six months to examine the effectiveness and safety of Amosartan Q tablet.

This study approved by the institutions' IRBs and was conducted in compliance with clinical research ethics regulations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hypertension and dyslipidemia
* Those who have already decided to administer Amosartan Q tablet under the medical judgment of the researcher
* Those who voluntarily decided to participate in this study and consented in writing to the consent form

Exclusion Criteria:

* Patients for whom use of Amosartan Q tablet is prohibited

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have hypertension and dyslipidemia
Sampling Method: Non-Probability Sample
Enrollment: 5400 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
percentage(%) of patients who achieved target blood pressure | 6 months
percentage(%) of patients who achieved target LDL-C | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hanmi Pharmaceutical Company Limited, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No